CLINICAL TRIAL: NCT00817193
Title: Early Screening and Exercise for Prevention of Disability in Persons Residing in Continuing Care Retirement Communities
Brief Title: Staying Healthy Through Education and Prevention Study
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LeadingAge (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHSA290200600024; 7581700 8-K72PS80 25505
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Disability
Keywords: Clinical trial; Short Physical Performance Battery; Disability; Senior Housing; Aging
MeSH Terms: interventions — Exercise; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Participants will begin to participate in walking sessions and strength building classes that will be offered at each location. Participants will be asked to attend a minimum of 1 strength class per week, with a target of doing 150 minutes of moderate exercise each week. The exercise classes will include stretching and counseling to help participants understand and address the barriers to becoming and staying involved in regular exercise.
  Interventions: Behavioral: Physical Activity
- Wellness (Active Comparator): Participants will begin to participate in a wellness program that will meet at each site twice per month. The first meeting will involve a lecture or presentation on a wellness-related topic. The second meeting will follow-up on concepts that were introduced in the first meeting, and will also to provide participants an opportunity to share experiences. Participants will be asked to attend both wellness sessions each month for whole year that the program is running.
  Interventions: Behavioral: Wellness

INTERVENTIONS:
Behavioral: Physical Activity — Physical Activity program
  Other Names: Exercise
  Arms: Physical Activity
Behavioral: Wellness — Wellness program
  Other Names: Active control
  Arms: Wellness

SUMMARY:
The purpose of this study is to test the effectiveness of a structured physical activity program, relative to a wellness program, in preventing the onset and progression of disability in the setting of senior housing communities, which are sometimes called housing with services.

DETAILED DESCRIPTION:
As the baby boom population ages, a large number of older adults have found that continuing care retirement communities (CCRCs) offer an attractive residential option. These communities include independent apartments, assisted living and skilled nursing options and often provide a menu of wellness services and a "safety net" of higher level care if/when that care is needed. CCRCs have proliferated in recent years and the number of older adults selecting this residential option is expected to continue. CCRCs represent a largely untapped provider setting in which interventions that have been proven effective in clinically-oriented, controlled studies of community-dwelling elderly can be translated into practice.

Multiple randomized studies have shown the benefits of physical activity interventions such as resistance and endurance exercises on a number of performance measures including walking speed, balance and ability to stand from a chair. These studies have shown that if given an exercise program matched to their needs, the onset and progression of disability can be decreased among persons who are identified at high risk of disability. However, most data supporting the beneficial effect of exercise in old age have been generated from studies conducted in highly controlled clinical trial settings, not in "real world" provider settings in which older adults live and function day-to-day. Thus, it is not known if screening for disability and implementing an exercise program among high risk elders can be effectively implemented in residential settings in a manner that not only promotes health and prevents disability, but that is also attractive to providers from a business standpoint and that can be incorporated into typical staffing patterns.

The American Association of Homes & Services for the Aging (AAHSA) is conducting a trial that builds on a strong evidence base of the beneficial effect of exercise in old age in an effort to accelerate translation of research into practice in CCRCs. The trial will screen CCRC residents for disability using a short set of performance measures called the Short Physical Performance Battery (SPPB). After identification of persons at risk for disability, we will enroll 320 CCRC residents to a program of moderate exercise or an active control arm focused on general wellness. The primary study endpoint is the SPPB score. Secondary endpoints include falls; hospitalizations, and death.

A key feature of the current proposal is that it seeks to extend findings from clinical studies into routine practice in the CCRC setting. This represents true translation of research into practice, and will offer providers an evidence base upon which to make informed decisions.

The trial will take place in 8 CCRCs operated by the Good Samaritan Society, the largest nonprofit provider of services to older adults in the country. Because of its large size and existing dissemination capacity, Good Samaritan is in a unique position to take a leadership role among aging services providers in terms of dissemination of effective, innovative programs in diverse residential settings, including CCRCs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Currently reside in independent or assisted living units of participating senior housing with services communities and intend to stay at facility without interruption for the next year
* Baseline SPPB scores between 3 and 9, inclusive.

Exclusion Criteria:

* Age < 65
* Severe cognitive impairment and/or inability to participate actively in the consent process (as determined by research staff).
* Myocardial infarction, stroke, hip fracture, hip or knee replacement, major heart surgery, including valve replacement or bypass surgery, or blood clot in leg or lungs in the previous 3 months.
* Self-reported inability to walk 13 feet with or without an assistive device
* Refusal to participate in the consenting process
* Failure to complete or attempt any of the 3 components of the SPPB for any non-physical reason
* SPPB scores less than 3 or more than 9.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery score | 12 months

SECONDARY OUTCOMES:
Incidence of Falls that result in participant being completely on the ground | 12
Incidence of hospitalization | 12 months
Incidence of Nursing home admission | 12 months
Incidence of emergence room visit | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helaine Resnick, PhD, Principal Investigator — LeadingAge
Locations (10):
- United States (10):
  - Good Samaritan Society - Mountain Home, Mountain Home, Arkansas
  - Good Samaritan Society - Loveland Village, Loveland, Colorado
  - Good Samaritan Society - Florida Luthern, DeLand, Florida
  - Good Samaritan Society - Kissemmee Village, Kissimmee, Florida
  - Good Samaritan Society - Cedar Lake Village, Olathe, Kansas
  - Good Samaritan Society - Westview Acres, Waconia, Minnesota
  - Good Samaritan Society - Hastings Village, Hastings, Nebraska
  - Good Samaritan Society - Manzano del Sol, Albuquerque, New Mexico
  - Good Samaritan Society - Fairlawn Village, Gresham, Oregon
  - Good Samaritan Society - Denton Village, Denton, Texas

REFERENCES:
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156